CLINICAL TRIAL: NCT04901520
Title: The Effects of Different Intensity Training on Dynamic and Static Balance of Elderly Women: A Randomized Controlled Trial
Brief Title: The Effects of Different Intensity Training on Dynamic and Static Balance of Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Kamran Hosseinzadeh Ghasemabad, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: A-GS47732
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Healthy Aging
Keywords: Older adults; Dynamic Balance; Static Balance; Resistance Training; High-Intensity training; Moderate-Intensity Training; Low-Intensity Training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: 3 intervention groups and one control group, assessed in 4 different times (baseline, 4th, 8th, and 12th weeks of intervention)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High Intensity Training (HIT) (Experimental): Participants trained at 80-90% of 1RM for 12 weeks, twice per week.
  Interventions: Other: High Intensity Training
- Moderate Intensity Training (MIT) (Experimental): Participants trained at 65-75% of 1RM for 12 weeks, twice per week.
  Interventions: Other: Moderate Intensity Training
- Low Intensity Training (LIT) (Experimental): Participants trained at 50-60% of 1RM for 12 weeks, twice per week.
  Interventions: Other: Low Intensity Training
- Control Group (CG) (No Intervention): Participants did not participate in any training and they advised to do their daily activity

INTERVENTIONS:
Other: High Intensity Training — High Intensity Training group performed resistance training with the intensity of 80 - 90 % of 1RM with 4 - 6 repetition
  Arms: High Intensity Training (HIT)
Other: Moderate Intensity Training — Moderate Intensity Training group performed resistance training with the intensity of 65 - 75 % of 1RM with 8 - 10 repetition
  Arms: Moderate Intensity Training (MIT)
Other: Low Intensity Training — Low Intensity Training group performed resistance training with the intensity of 50 - 60 % of 1RM with 12 - 14 repetition
  Arms: Low Intensity Training (LIT)

SUMMARY:
In this study, investigators tried to find a useful and safe way of training for the elderly population which can help this population to improve their fitness factors as fast as possible. investigators have tried to see if different intensity training has different effects on the dynamic and static balance of elderly women in different time points (4, 8, and 12 weeks). Investigators hypothesized that Higher intensity would be more effective to improve balance at different time points. The participants were trained twice per week and each session contain 4 exercises ( leg press, leg extension, leg curl, and seated calf raises) and the data have been collected at the pre-test and 4th, 8th, and 12th weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years old and above.
* Orientation to place, time, and person, able to follow the simple instructions, and perform the exercises.
* Without any health problems that would interfere with their safety or ability to complete high and low-intensity training such as the occurrence of myocardial infarction in the past six months, recent heart attack, uncontrolled hypertension (Blood Pressure >166/96 mm Hg), a broken leg in the past six months, diagnosed osteoporosis, and diagnosed stage three and four of heart failure.

Exclusion Criteria:

* Participation in regular balance or lower body resistance training during the past three months (at least twice per week).
* The health issues that might confound the study results, including lower- body neuropathy, stroke within the past year, Parkinson's disease, diagnosed vestibular disorders, severe vision (self-rated vision as poor or very poor even when wearing glasses or contact lenses), and lower- extremity joint replacements.
* Taking the regular medication's impairing balance ability (Antidepressants, Neuroleptics or Benzodiazepines) or muscle strength (Corticosteroids).
* Elderly with dementia

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Mean of Front Reach Test at 4, 8, and 12 weeks | Baseline, 4th weeks, 8th weeks, 12th weeks
  The distance that subject can lean forward measured in centimetre (cm) with measuring tape. The higher score is better. The minimum is 5 cm and maximum 50 cm
Change from Baseline in the Mean of Lateral Reach Test at 4, 8, and 12 weeks | Baseline, 4th weeks, 8th weeks, 12th weeks
  The distance that subject can lean to the side measured in centimetre (cm) with measuring tape. The higher score is better. Minimum is 5 cm and maximum is 50 cm
Change from Baseline in the Mean of One Leg Stand at 4, 8, and 12 weeks | Baseline, 4th weeks, 8th weeks, 12th weeks
  The timed that subject can stand in 1 leg recorded in second using a stop watch. The higher score is better. minimum is 1 second and maximum is 30 second
Change from Baseline in the Mean of Tandem Stand Test at 4, 8, and 12 weeks | Baseline, 4th weeks, 8th weeks, 12th weeks
  The timed that subject can stand one leg front and one leg back condition recorded in second using a stop watch. The higher score is better. Minimum is 1 second and maximum is 30 second

CONTACTS AND LOCATIONS:
Locations (1):
- Fit House Bukit Rimao, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided